CLINICAL TRIAL: NCT06182969
Title: A Randomized, Double-blind, Placebo-controlled Phase I/II Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of APG-2575 in Patients With Mild-to-moderate Systemic Lupus Erythematosus.
Brief Title: A Study of APG-2575 in Patients With Mild-to-moderate Systemic Lupus Erythematosus.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Collaborators: Suzhou Yasheng Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APG2575SC101
Record Dates: First submitted 2023-12-03; First posted 2023-12-27 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: SLE
Keywords: SLE; APG-2575
MeSH Terms: interventions — Lisaftoclax

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APG-2575 (Experimental): Dose escalation
  Interventions: Drug: APG-2575
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: APG-2575 — Take orally once daily (QD) for 12 weeks.
  Arms: APG-2575
Other: Placebo — Take orally once daily (QD) for 12 weeks.
  Arms: Placebo

SUMMARY:
To evaluate the safety, tolerability, pharmacokinetics and pharmacokinetics of multi-dose APG-2575 in mild-to-moderate systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled Phase I/II study. About 40 participants will be recruited to receive either APG-2575 or a placebo, with doses from 200mg up to 800mg.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosis of systemic lupus erythematosus for at least 6 months.
* 2. On stable treatment for systemic lupus erythematosus before first dose at least 28 days.
* 3. SLEDIA-2000 score: 4-12
* 4.Other than systemic lupus erythematosus, subject should be in general good health.

Exclusion Criteria:

* 1. Severe systemic lupus erythematosus.
* 2. Significant autoimmune disease other than lupus.
* 3. Significant, uncontrolled or unstable disease in any organ.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. | Up to 1 year
  According to CTCAE v5.0, the number and frequency of adverse events of test drug were assessed.

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of APG-2575 in SLE patients. | At Day1 and Day 28 since the first dose of study drug.
  To evaluate the metabolic characteristics of APG-2575 in SLE patients
Area under the plasma concentration versus time curve (AUC) of APG-2575 in SLE patients. | At Day1 and Day 28 since the first dose of study drug.
  To evaluate the metabolic characteristics of APG-2575 in SLE patients
Time to Peak (Tmax) of APG-2575 in SLE patients. | At Day1 and Day 28 since the first dose of study drug.
  To evaluate the metabolic characteristics of APG-2575 in SLE patients
Assessment of SLE disease activity using SLEDAI（Systemic Lupus Erythematosus Disease Activity Index）-2000. | Up to 1 year
  To evaluate the patients' efficacy.

OTHER OUTCOMES:
Change in the number and percentages of immune cells clusters. | Up to 1 year
  The changes of immune cell clusters from baseline.
Change in the number and percentages of cytokines. | Up to 1 year
  The changes of cytokines from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Chen, Ph.D, Principal Investigator — Renji Hospital Shanghai Jiaotong University School of Medical
Locations (1):
- Renji Hospital Shanghai Jiaotong University School of Medical, Shanghai, Shanghai Municipality, China